CLINICAL TRIAL: NCT07284082
Title: The Synergistic Effects of Menopause and HIV on Cardiovascular Disease Risk in Women
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 25-43802; K23HL178394 (NIH)
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: HIV; Menopause; Cardiovascular (CV) Risk; Carotid Arteriosclerosis; Body Composition
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MACS-WIHS Combined Cohort Study
  Interventions: Diagnostic Test: Whole body MRI

INTERVENTIONS:
Diagnostic Test: Whole body MRI — Whole body MRI will be performed as part of a study protocol

SUMMARY:
Menopause is associated with the acceleration of many comorbidities, including cardiovascular disease. Whether HIV and menopause together increase cardiovascular disease risk is a key knowledge gap. The goal of this observational study is to address this knowledge gap by looking at the role of menopause on cardiovascular disease risk factors such as insulin resistance, hypertension, hyperlipidemia, and carotid atherosclerosis using previously collected data. The investigators will look at underlying causes for cardiovascular diseases worsening in menopausal women with HIV by looking at the role of increased inflammation in the body and whether this is altered by weight. The investigators achieve this by enrolling participants who are willing to undergo a whole body MRI.

ELIGIBILITY:
Inclusion Criteria:

* 90 non-pregnant women with HIV (approximately 30 in each menopausal phase) from the San Francisco MWCCS site.

Exclusion Criteria:

* Women who are not virally suppressed (HIV RNA >200 copies/mL)
* Women who are not on antiretroviral therapy
* Women who have a history of hysterectomy or oophorectomy
* Women who are receiving treatment for active cancer or tuberculosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with HIV who are enrolled in the MWCCS.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Markers of immune activation and inflammation | These markers will be measured from blood work collected at the scheduled study visit [Day 1] close to the time of MRI and thus will be collected at only one time point.
  sCD14 (monocyte activation), sCD163 (M2 macrophage activation), CRP (inflammation), IL-6 (inflammation), IP-10 (interferon-inducible protein), TNFα (inflammation), MCP-1 (inflammation), sTNFRI & RII (inflammation). There are no units as they will be normalized based upon their interquartile range.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Abelman, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No